CLINICAL TRIAL: NCT02592239
Title: Hedonic Perception and Brain Activity Response to Meal in Health and Functional Dyspepsia
Brief Title: Hedonic Perception and Brain Activity Response to Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AG)214/2012 Addendum
Record Dates: First submitted 2015-03-17; First posted 2015-10-30 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2016-09

CONDITIONS: Dyspepsia
Keywords: Functional brain MRI; functional dyspepsia; hedonic response
MeSH Terms: conditions — Dyspepsia | interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Functional dyspepsia patients will be studied using functional brain MRI before and after receiving a test meal. Cognitive and hedonic response will be evaluated using 10 score scales.
  Interventions: Device: Functional brain MRI; Dietary Supplement: A warm ham and cheese sandwich and a 200 ml fruit juice
- Controls (Experimental): Healthy subjects recruited by public advertisement will be studied using functional brain MRI before and after receiving a test meal. Cognitive and hedonic response will be evaluated using 10 score scales.
  Interventions: Device: Functional brain MRI; Dietary Supplement: A warm ham and cheese sandwich and a 200 ml fruit juice

INTERVENTIONS:
Device: Functional brain MRI — Functional brain MRI before and after test meal ingestion
Dietary Supplement: A warm ham and cheese sandwich and a 200 ml fruit juice

SUMMARY:
The purpose of this study is to determine the relationship between brain activity and the perception of subjective hedonic sensations in response to a meal using functional MRI.

DETAILED DESCRIPTION:
Functional MRI brain imaging will be performed in patients with functional dyspepsia and healthy controls in basal conditions and after a palatable test meal. During the study, the cognitive response and the hedonic dimension will be measured using 10 score scales.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 yrs
2. Body mass index between 18-30 Kg/m2
3. Right-handed

Exclusion Criteria:

1. Subjects with clinical history of eating-disorders
2. Subjects with clinical history of significant head-trauma
3. Subjects with known serious illness: clinically significant cardiac, vascular, liver, pulmonary, or psychiatric disorders (as evaluated by the Investigator).
4. Subjects with a known history of alcohol or drug abuse in the previous 6 months.
5. Subjects using medications with SNS effects that cannot be discontinued, such as: antidepressants, pregabalin, gabapentin.
6. Women that are pregnant or that are breast-feeding.
7. Claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in activity in specific brain regions measured by functional MRI | 3 hours
  To determine the brain response to a meal in patients with functional dyspepsia and healthy subjects.
Cognitive and hedonic perception measured on 10 score scales (composite outcome) | 3 hours
  To determine the cognitive and hedonic response to a meal in patients with functional dyspepsia and healthy subjects.

SECONDARY OUTCOMES:
Metabolomic response measured in serum by NMR spectroscopy | 3 hours
  To identify the metabolomic substrate of the cognitive and brain responses to a meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Research Institute, Barcelona, Spain

REFERENCES:
- [Background] Malagelada C, Accarino A, Molne L, Mendez S, Campos E, Gonzalez A, Malagelada JR, Azpiroz F. Digestive, cognitive and hedonic responses to a meal. Neurogastroenterol Motil. 2015 Mar;27(3):389-96. doi: 10.1111/nmo.12504. Epub 2015 Jan 3. PMID 25557693
- [Background] Liu P, Qin W, Wang J, Zeng F, Zhou G, Wen H, von Deneen KM, Liang F, Gong Q, Tian J. Identifying neural patterns of functional dyspepsia using multivariate pattern analysis: a resting-state FMRI study. PLoS One. 2013 Jul 12;8(7):e68205. doi: 10.1371/journal.pone.0068205. Print 2013. PMID 23874543
- [Background] Zeng F, Qin W, Liang F, Liu J, Tang Y, Liu X, Yuan K, Yu S, Song W, Liu M, Lan L, Gao X, Liu Y, Tian J. Abnormal resting brain activity in patients with functional dyspepsia is related to symptom severity. Gastroenterology. 2011 Aug;141(2):499-506. doi: 10.1053/j.gastro.2011.05.003. Epub 2011 May 17. PMID 21684280
- [Background] Van Oudenhove L, Vandenberghe J, Dupont P, Geeraerts B, Vos R, Dirix S, Bormans G, Vanderghinste D, Van Laere K, Demyttenaere K, Fischler B, Tack J. Abnormal regional brain activity during rest and (anticipated) gastric distension in functional dyspepsia and the role of anxiety: a H(2)(15)O-PET study. Am J Gastroenterol. 2010 Apr;105(4):913-24. doi: 10.1038/ajg.2010.39. Epub 2010 Feb 16. PMID 20160711